CLINICAL TRIAL: NCT04143165
Title: Ultrasound Guided Epidural Block in Axial SPA Patient With Limited Spine Mobility: a Prospective Pilot Randomized Controlled Trial
Brief Title: Ultrasound Guided Epidural Block in Axial SPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous, Associate professor, Sohag University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20/10/2019
Record Dates: First submitted 2019-10-26; First posted 2019-10-29 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Epidural Block in Axial Spondyloarthritis
MeSH Terms: interventions — Anesthesia, Epidural; Lidocaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural block (Active Comparator): Group I patients received caudal epidural injections with 1% lidocaine hydrochloride (xylocaine Astra Zeneca) 9 mL mixed with 1 mL of triamcinolone 40 milligrams (Kenacort Bristol Myers Squip)
  Interventions: Drug: Epidural block with lidocaine and triamcinilone
- control group (No Intervention): patients did not receive injection

INTERVENTIONS:
Drug: Epidural block with lidocaine and triamcinilone — caudal epidural injections with 1% lidocaine hydrochloride (xylocaine AstraZeneca) 9 mL mixed with 1 mL of triamcinolone 40 milligrams (Kenacort Bristol Myers Squip)
  Arms: Epidural block

SUMMARY:
Study Design: A randomized, prospective, pilot, controlled trial. Setting: Rheumatology and rehabilitation department Minia University and Sohag University Objectives: To evaluate the effectiveness of caudal epidural injections with triamcinolone and lidocaine in managing limited spine mobility in axial SPA.

Methods: Patients were randomly assigned to one of 2 groups, Group I patients received caudal epidural injections with 1% lidocaine hydrochloride (xylocaine AstraZeneca) 9 mL mixed with 1 mL of triamcinolone 40 milligrams (Kenacort Bristol Myers Squip), whereas Group II patients did not receive. Both groups were age and sex matched and both were under treatment with anti TNF and NSAIDs with or without sDMARDs.

ELIGIBILITY:
Inclusion Criteria:

* all participants fulfilled the ASAS criteria for axial SPA
* all participants under treatment including bDMARDS and sDMARDs beside NSAIDs

Exclusion Criteria:

* Naive patients not under treatment
* limitation of spine flexion due to non inflammatory causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
change in pain | Baseline, after 2 weeks and after 8 weeks
  visual analogue scale for pain minimum score 0 maximum score 10
Change in functional ability of the patient | Baseline, after 2 weeks and after 8 weeks
  Bath Ankylosing Spondylitis Functional Index (BASFI) minimum score 0 maximum 100, Oswestry Disability Index (ODI) minimum 0 no disability, maximum 100 means complete disability
Change in spinal mobility | Baseline, after 2 weeks and after 8 weeks
  Bath AS Metrology Index (BASMI) minimum score 0 maximum 50, modified Schober test less than 5 cm yield means limited mobility, Lateral lumbar flexion more than 55 cm yield means limited lateral flexion
Change in ASDAS- CRP score | Baseline, after 2 weeks and after 8 weeks
  ≥ 1.1 reduction in the initial score, less than 1.3 inactive disease, between 1.3 and 2.1 moderate, between 2.1-3.5 high disease activity, > 3.5 very high disease activty

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No
The consent form does not include this item

REFERENCES:
- [Derived] Elsaman AM, Hamed A, Radwan AR. Ultrasound-guided epidural block in axial spondyloarthritis patients with limited spine mobility: a randomized controlled trial. Korean J Pain. 2021 Jan 1;34(1):114-123. doi: 10.3344/kjp.2021.34.1.114. PMID 33380574